CLINICAL TRIAL: NCT04748289
Title: Integrated Platform for Multimodal Patient Monitoring and Therapy Support in ICU Patients: Interventional Study With First ICU Cockpit Software Applications
Brief Title: ICU Cockpit Apps: Interventional Study With First ICU Cockpit Software Applications
Acronym: ICUCockpiApp
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasilibilty
Sponsor: Emanuela Keller (Other)
Responsible Party: Sponsor-Investigator, Emanuela Keller, Neurocritical Care Unit, University Hospital Zurich, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-02177
Record Dates: First submitted 2021-01-27; First posted 2021-02-10 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Clinical Decision Support System
Keywords: Secondary brain injuries; COVID-19; Subarachnoid hemorrhage
MeSH Terms: conditions — COVID-19; Subarachnoid Hemorrhage

STUDY DESIGN:
Intervention Model Description: Open labelled, single centre clinical investigation, with the new ICU Cockpit Software Platform (medical device).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NICU patients (Experimental): All patients admitted to the Neurointensive Care Unit (NICU)
  Interventions: Device: ICU Cockpit software testing

INTERVENTIONS:
Device: ICU Cockpit software testing — the ICU Cockpit Software Platform is intended to be used for monitoring of patient characteristics and vital physiological parameters in patients at the Neurointensive Care Unit of the University Hospital Zurich.
  Furthermore, three different applications for prognostication and prediction of complications will be tested:
  1. ICU Cockpit COVID-19 for remote monitoring of isolated patients,
  2. ICU Cockpit Stable State for a comprehensive visualization of vital parameters and as additional aid in early detection of imminent critical complications
  3. ICU Cockpit Cerebral Ischemia for the prediction of delayed DCI in patients with subarachnoid hemorrhage (SAH).

SUMMARY:
In neurocritical care, besides the standard intensive care monitoring, even more data are obtained from the very complex pathophysiological changes in brain disease. Medical staff for decision-making cannot integrate the huge amount of clinical data generated every second and visualized on different monitors, anymore. Lack of data integration and usability is a major reason that only few of the knowledge physicians use in this field is evidence based.

Early warning systems, powered by predictive algorithms that detect critical states before they happen would allow the staﬀ to intervene early and mitigate or even prevent such a critical state.

DETAILED DESCRIPTION:
Background:

Since 2014, the project "ICU-Cockpit" has been set up at the Neurointensive Unit of the University Hospital Zurich in collaboration with the University of Zurich and ETH Zurich. State-of-the-art information technology collects, synchronizes and encrypts data from numerous medical devices in real time. The project is aimed at initiating a fundamental development in emergency and intensive medicine - and bringing about a substantial improvement in the way diagnostics, treatment and risk management are handled in everyday clinical practice.

Based on video monitoring, algorithms for early alarm systems and therapy support have been already developed. In order to make the algorithms usable for clinical practice, a user interface (GUI) is currently being developed in cooperation with the University of Applied Sciences Northwestern Switzerland (FHNW), see appendix 15. The GUI allows to visualize and interpret the multimodal patient data in a comprehensive manner.

In 2016, a research project started at the NICU of the University Hospital Zurich started with the title "ICU Cockpit: Integrated platform for multimodal patient monitoring and therapy support in neurocritical care" (BASEC No. 2016-01101). The purpose of the single site project is to set up an integrated platform (scientific prototype of ICU Cockpit software platform) for multimodal patient monitoring and therapy support in neurocritical care, and as a second step to develop and validate algorithms for some first clinical applications. Furthermore, automatic artefacts detections (i.e., number of false and true alarms in ICU Cockpit in comparison to standard monitoring system) are assessed and algorithms are developed for the early detection of epileptic seizures and secondary impairment of cerebral perfusion.

The objective of this current clinical investigation is the verification and validation of the ICU Cockpit software platform and the following three different applications for prognostication and prediction of complications:

a) ICU Cockpit COVID-19 for remote monitoring of isolated patients, b) ICU Cockpit Stable State for a comprehensive visualization of vital parameters and as additional aid in early detection of imminent critical complications c) ICU Cockpit Cerebral Ischemia for the prediction of delayed cerebral ischemia in patients with subarachnoid hemorrhage (SAH).

1. ICU Cockpit COVID-19 for remote monitoring of isolated patients Having infected more than 100 000 people in 100 countries, the coronavirus disease 2019 (COVID-19) has become a pandemic. In China, up to 10% of patients with COVID-19 became severely ill requiring intensive care treatment mostly due to pneumonia, acute respiratory distress syndrome (ARDS) and multiorgan failure. In Italy, having about 5200 beds in intensive care units (ICUs), already 1028 were already devoted to patients with COVID-19 by March 11. Furthermore, 20% of health-care professionals, at this time, have become already infected, and some have died. For the United States, without self-isolation and for R0 = 2 and R0 = 2.5, respectively, ICU admissions are projected to become 17.4 to 25.7 per 1,000 population, which would significantly exceed the capacity of the existing 100,000 ICU beds in the US. Also, in Switzerland the health care system and especially ICUs are facing extraordinary challenges as human resources for ICU professionals are limited.

   Advances in medical informatics have the potential to facilitate medical care and save personnel resources not only in the ambulatory sector but in the ICUs especially during epidemics. In intensive and emergency medicine, the situation is compounded by real-time signals from multiple sensors on, as well as inside the human body. In an emergency situation, in particular, it is not possible to integrate this flood of information rapidly into the decision-making process.

   Remote monitoring of strictly isolated patients especially reduces routes and walking of the staff, the number of close contacts with infected patients and therefore, virus transmission. The safety of patients will be increased by a reduction of stress and burnouts in nurses and medical doctors, which often work in crisis over time.
2. ICU Cockpit Stable State As a first application a software called "stable state" has been developed recently. Vital parameters as arterial blood pressure, intracranial pressure and many others are hard to read in a glance due to their high information density. Since the human body is a complexly inter-connected system, these biosignals are also heavily correlated. Experienced clinicians can recognize deviations in the correlational structure of several signals, but it is impossible to grasp the full picture for the huge amount of available data. However, subtle correlational changes may indicate an instable state of a patient before these changes are visible in a specific signal or its compound measure.

   An algorithm which computes the inter-dependencies in an arbitrary set of signals during a stable phase of the patient was recently developed. This stable state is compared to an on-line estimate of the current state. Correlational changes are didactically reduced and visualized in a Mondrian-like display for quick comparisons of current and past states.

   The application "stable state" as part of the GUI ICU Cockpit is planned to be implemented as an additional aid in early detection of imminent critical complications.
3. ICU Cockpit Cerebral Ischemia Cerebral vasospasm (CVS) is a delayed morphologic narrowing of cerebral arteries, occurring 4 to 10 days after aneurysmal subarachnoid hemorrhage. Classically, CVS has been associated with delayed cerebral ischemia (DCI), which ultimately leads to cerebral infarction associated with morbidity and mortality. This has been sort of a paradigm, and the term CVS has been often misused to describe clinical signs of DCI. The majority of research was focused on the assumption CVS to be solely responsible for DCI. Today, it is well accepted that not all patients with CVS develop DCI. Inversely, DCI can occur in the absence of CVS. Recent review of the literature indicates that CVS is not the only cause of DCI and that the entire picture of DCI is multifactorial. There is an ongoing debate about this issue, however cerebral infarction on imaging studies might be the most appropriate measure of DCI beside functional outcome. Therefore, an algorithm to predict DCI based on a random forest model has been developed, which allows to identify biomarkers for the occurrence 24h to 48 hours before.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the Neurointensive Care Unit (NICU)
* Informed Consent by signature from representative / patient

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Verification of ICU Cockpit software for remote monitoring of isolated patients | 2 years
  Repeatability, reliability, performance of prediction of models results will be testet against ground truth (annotations by experts).
Verification of ICU Cockpit software ICU Cockpit Stable State | 2 years
  Repeatability, reliability, performance of prediction of models results will be testet against ground truth (annotations by experts).
Verification of ICU Cockpit software Cerebral Ischemia | 2 years
  Prediction score estimated by the app ICU Cockpit Cerebral Ischemia compared to probability estimation by medical experts in surveys.
Adverse events, complaints and use-errors reporting | 2 years
  Reporting of adverse events (incl. device deficiencies), complaints as well as use-errors.
Usability testing | 2 years
  Usability testing by distributing the Software Usability Questionnaire to involved medical staff (n=65).

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Keller, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Callaway E, Cyranoski D, Mallapaty S, Stoye E, Tollefson J. The coronavirus pandemic in five powerful charts. Nature. 2020 Mar;579(7800):482-483. doi: 10.1038/d41586-020-00758-2. No abstract available. PMID 32203366
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Hollander JE, Carr BG. Virtually Perfect? Telemedicine for Covid-19. N Engl J Med. 2020 Apr 30;382(18):1679-1681. doi: 10.1056/NEJMp2003539. Epub 2020 Mar 11. No abstract available. PMID 32160451
- [Background] Vergouwen MD, Ilodigwe D, Macdonald RL. Cerebral infarction after subarachnoid hemorrhage contributes to poor outcome by vasospasm-dependent and -independent effects. Stroke. 2011 Apr;42(4):924-9. doi: 10.1161/STROKEAHA.110.597914. Epub 2011 Feb 10. PMID 21311062